CLINICAL TRIAL: NCT04577586
Title: Negative Oral Contrast Agents Utilization in PET/CT Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nahla Mostafa Mahmoud Bashank, PhD, Assiut University
Other Study IDs: Negative oral contrast PET/CT
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: PET/CT; Oral Contrast
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Water: Patients who ingested only water as an oral contrast
  Interventions: Other: oral contrast
- Milk: Patients who ingested milk as an oral contrast
  Interventions: Other: oral contrast
- Mannitol: Patients who ingested mannitol as an oral contrast
  Interventions: Other: oral contrast

INTERVENTIONS:
Other: oral contrast — negative oral contrast utilization in PET/CT studies

SUMMARY:
To compare the performance of different negative oral contrast agents in bowel distension in patient referred for PET/CT studies for various causes aiming for identification of ideal oral contrast agent(OCA).

DETAILED DESCRIPTION:
Evaluation of gastrointestinal pathology depends on adequate bowel distention, which optimizes resolution of the bowel wall and contents. Traditionally, high-attenuation oral Contrast material in the form of iodine solutions or barium suspensions has been used to obtain bowel distension in MDCT examinations

Traditional high-contrast oral agents like iodine solutions, and barium suspensions which due to overcorrection problems in PET-CT interpretation lowers the accuracy of diagnosis. Negative oral contrast agents like water, air, fat containing agents used with 12.5% corn oil and polyethylene glycol has been used in radiological studies. Milk with 4% fat content has also been tested out in radiological studies and found to be effective. As it is more easily available, palatable, and acceptable especially, by children it needed to be tested in the visualization of the GIT in the PET-CT studies compared to other negative contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to our unit for PET/CT study for various causes

Exclusion Criteria:

* Patients with GIT disease.
* Pregnancy and lactation.
* Severely ill patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients in our institution who prepared for PET-CT with administration of oral contrast material
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
compare the performance of different negative oral contrast agents in PET/Ct studies | baseline
  comparing the effect of different oral contrast on bowel distention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer SA, Gawde S. Utility of negative oral contrast (milk with 4% fat) in PET-CT studies. Indian J Nucl Med. 2012 Jul;27(3):151-5. doi: 10.4103/0972-3919.112719. PMID 23919067
- [Background] Koo CW, Shah-Patel LR, Baer JW, Frager DH. Cost-effectiveness and patient tolerance of low-attenuation oral contrast material: milk versus VoLumen. AJR Am J Roentgenol. 2008 May;190(5):1307-13. doi: 10.2214/AJR.07.3193. PMID 18430848